CLINICAL TRIAL: NCT01302444
Title: Randomized Placebo Controlled Trial of Treprostinil Infusion Combined With Oral Tadalafil or Placebo in Pulmonary Arterial Hypertension
Brief Title: Treprostinil Combined With Tadalafil for Pulmonary Hypertension
Acronym: T2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: One subject enrolled and completed this study. The study was stopped due to poor recruitment.
Sponsor: Rhode Island Hospital (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T2 Trial
Record Dates: First submitted 2011-02-16; First posted 2011-02-24 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2012-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: treprostinil; pulmonary hypertension, tadalafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Tadalafil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator): first 4 weeks are for adjusting treprostinil dose, then Tadalafil 40mg daily for 12 weeks, Group is randomly chosen from entire cohort
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): first 4 weeks for adjusting treprostinil dose, then Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil 40mg for 12 weeks
  Other Names: Adcirca
  Arms: Tadalafil
Drug: Placebo — Placebo for 12 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Objectives: To test whether the combined administration of the medications treprostinil(a prostacycline therapy), and tadalafil(a PDE-5 [ phosphodiesterase type 5]Inhibitor therapy) is better than the administration of treprostinil alone. This treatment would be offered to newly diagnosed patients with pulmonary arterial hypertension who are on no treatment for this disease and are deemed candidates for the medication treprostinil by their physician. The combination therapy will be compared to single therapy with only treprostinil in a double-blind manner.

Current therapy is to begin one treatment, either a PDE5 inhibitor or a prostacycline, depending on the severity of the patient's PAH (pulmonary arterial hypertension) disease and add additional therapies as deterioration occurs. This treatment could add two agents initially.

Secondary objectives are: To improve pulmonary arterial pressures as measured through a cardiac echocardiogram, improve the subject's 6minute walk distance, delaying the time to clinical worsening, and lowering plasma BNP levels.

Research Procedures: To begin the administration of both treatments at the same time.

Time period is 16 weeks with a one- year follow-up. Cardiac Echocardiograms, clinic physician exams, and lab work will be followed. Subjects will be between the ages of 18 - 75.

DETAILED DESCRIPTION:
Background: Many cardiovascular diseases such as essential hypertension, coronary artery disease and congestive heart failure respond better to combinations of vasoactive drugs, than to therapy with a single agent. Three categories of pulmonary anti-hypertensive medications have been developed over the last 20 years, but their effect on management of PAH when used in combination are mostly unknown. Two of the pulmonary arterial hypertension (PAH) drug groups are prostacyclines, and PDE5 inhibitors. Although the effects of prostacyclins are mediated via cAMP (cyclic guanosine monophosphate) and the effects of PDE5 inhibitors are mediated via cGMP, there is considerable cross talk between these nucleotides suggesting that adequate levels of both may be needed to maintain normal pulmonary vascular tone and cellular growth responses.

Objective/Hypothesis: This proposal hypothesizes that increasing the levels of both nucleotides (prostacyclines and PDE5 inhibitors), may be more efficacious in the treatment of PAH than increasing either one alone.

Specific Aims: The primary objective of this study is to determine if the combination of treprostinil infusion combined with tadalafil is more efficacious than treprostinil alone in improving the change from baseline in the 6 minute walking distance after 16 weeks of therapy.

Study Design: The proposed study is a multi-center, randomized, double blind, two cohort, parallel group, and 16-week study with 1-year long-term follow-up. The study aims to compare the efficacy of combination therapy with treprostinil infusion and tadalafil to treprostinil infusion alone.

Study Population: All patients who have been newly diagnosed with PAH and who, after consultation with their physician, have elected to be treated with treprostinil infusion will be invited to participate. A total of 66 subjects will be sort to enroll.

Treprostinil dosing will follow a 4 week up-titration schedule with a target 4week dose of 8ng/kg/min minimum, followed by a 12 week randomized tadalafil period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18-80 years of age
2. World Health Organization Group 1 PAH

   1. Idiopathic PAH
   2. Heritable PAH
   3. PAH associated with connective tissue disease
   4. PAH associated with surgical repair of congenital left to right shunt
   5. PAH associated with anorectic drug use
3. WHO functional Class III-IV
4. 6 minute walking distance > 150-meters and < 450 meters
5. Right heart catheterization showing mean PAP (pulmonary arterial pressure)> 25 mmHg and PCWP (pulmonary capillary wedge pressure) < 15 mmHg within 6 months of study entry.

Exclusion Criteria:

1. Pulmonary hypertension associated with

   a. Portal hypertension b. HIV infection c. Pulmonary venous hypertension defined as PCWP > 15 mmHg d. Chronic lung disease defined as i. FEV1(forced expiratory volume at one second

   )/FVC (forced vital capacity) less than 0.65 ii. TLC < 0.70 iii. Untreated Sleep Apnea with AHI (apnea-hypopnea index )> 20 or hemoglobin oxygen saturation nadir < 87% e. Chronic Thromboembolic Disease f. Sarcoidosis g. Pulmonary veno occlusive disease (PVOD)
2. Concomitant use of nitrates (any form) either regularly or intermittently.
3. Concomitant use of potent CYP3A inhibitors (e.g., ritonavir, ketoconazole, itraconazole)
4. Vascular disease of the retina including retinitis pigmentosa, any sudden vision loss, including any damage to the optic nerve or NAION
5. low blood pressure or high blood pressure that is not controlled
6. Postural hypotension
7. Inability to manage home infusion therapy
8. Pulmonary vasodilator therapy with any phosphodiesterase inhibitor or endothelin receptor antagonist within 30 days of study entry
9. Participation in a clinical investigational study within previous 30 days
10. Renal failure defined as:

    1. estimated creatinine clearance < 30 ml/min
    2. serum creatinine > 2.5 mg/dl
11. Subjects with liver function abnormalities (ALT [Alanine Aminotransferase or AST (Alanine Aminotransferase ) > 3 times the upper limit of normal at screening or at baseline) or chronic liver disease
12. History of hypersensitivity reaction or adverse effect related to tadalafil
13. Life expectancy < 12 months
14. History of deformed penis shape, an erection that lasted more than 4 hours, or Peyronie's disease.
15. Blood cell problems such as sickle cell anemia, multiple myeloma, or leukemia
16. Pregnant or planning to become pregnant or breast feed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Klinger, MD, Study Director — Rhode Island Hospital
Locations (9):
- United States (9):
  - Maine Medical Center, Portland, Maine
  - Tuft's New England Medical Center, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Saint Barnabas Health Care System, Newark Beth Israel Medical Center, Newark, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- See also: treprostinil — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2515411/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Time Frame: 16 weeks
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Adverse Events Are no Greater Than With Treprostinil Infusion Alone
Time Frame: 16 weeks
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: WHO Functional Class Will Improve or Remain Stable
Time Frame: 16 weeks
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Hospitalizations
Time Frame: 16 weeks
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 6 Minute Walking Distance Change Will Improve
Time Frame: 16 weeks of therapy
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Tei Index Change by Transthoracic Echocardiography
Time Frame: 16 weeks of therapy
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma BNP (Brain Natriuretic Peptide)Level Change
Time Frame: 16 weeks of therapy
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Pulmonary Arterial Systolic Pressure (PASP)as Assessed by Transthoracic Echocardiography Using Doppler Ultrasound
Time Frame: 16 weeks
Population: data not reported for one participant for anonymity
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No